CLINICAL TRIAL: NCT01428648
Title: Impact of Dance Therapy on Parkinson's Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment slow
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 133272
Record Dates: First submitted 2011-09-02; First posted 2011-09-05 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Parkinson's Disease
Keywords: Parkinson; ballroom dancing
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Active Comparator): group of patients receiving ballroom dancing classes
  Interventions: Behavioral: Ballroom Dancing Classes
- control (No Intervention): group of patients who will not receive dancing classes.

INTERVENTIONS:
Behavioral: Ballroom Dancing Classes — bi-weekly, 12-Week ballroom dance classes
  Arms: intervention

SUMMARY:
Parkinson's disease (PD) affects ability of individuals to perform unconscious learned motor tasks, affects quality of life and has been associated with depression. The purpose of this study is to investigate the effect of dance therapy on motor performance, quality of life and depression in PD patients, by comparing certain symptoms between a group of subjects with PD who undergo ballroom dancing classes and a control group of subjects with PD. The investigators will assess mental status, severity of PD, quality of life and depression using rating scales. Subjects will be randomized to intervention and control group. Intervention group will participate in dance therapy for 12 weeks and will be examined at 12 and 20 weeks. Control group will be examined at same time intervals. Classes will follow a curriculum designed by Arthur Murray Dance Studio Staff. The investigators do not anticipate significant risk for participants.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older, both males and females, all races and all ethnicities
* Idiopathic Parkinson's disease diagnosed using United Kingdom Parkinson's Disease Society brain bank diagnostic criteria
* Mild to moderate disease severity (Stage 2 to 3 on the Modified Hoehn and Yahr scale)
* Stable medication regimen for a minimum of 1 month before testing
* Ability to ambulate independently without using a walking aid
* Ability to give informed consent

Exclusion Criteria:

* Prior enrollment in a dancing class during the last 6 months
* Presence of another neurological or medical disorder likely to affect gait or causing frequent falls (rheumatologic/orthopedic disease, stroke, myelopathy, severe neuropathy)
* Significant cognitive decline (MMSE ≤ 24)
* Visual deficit
* Hearing deficit that impairs music perception
* Psychotic symptoms
* Symptomatic heart disease
* Depression associated with suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Effect of ballroom dancing classes on motor function in patients with Parkinson's disease. | 3 and 5 months
  The improvement in participant's motor function will be measured by the UPRS III score. The aim is to detect an 18-20% difference in UPDRS III scores among the two groups.

SECONDARY OUTCOMES:
Effect of ballroom dancing classes on depression in patients with Parkinson's disease. | 3 and 5 months
  The improvement in participant's depression will be measured by the Hamilton Depression Scale.
Effect of ballroom dancing classes on quality of life of patients with Parkinson's disease. | 3 and 5 months
  The improvement in participant's quality of life will be measured by the Parkinson's Disease-39 questionnaire PDQ-39 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Maalouf, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Background] Gelb DJ, Oliver E, Gilman S. Diagnostic criteria for Parkinson disease. Arch Neurol. 1999 Jan;56(1):33-9. doi: 10.1001/archneur.56.1.33. PMID 9923759
- [Background] Park A, Stacy M. Non-motor symptoms in Parkinson's disease. J Neurol. 2009 Aug;256 Suppl 3:293-8. doi: 10.1007/s00415-009-5240-1. PMID 19711119
- [Background] Ransmayr G. Physical, occupational, speech and swallowing therapies and physical exercise in Parkinson's disease. J Neural Transm (Vienna). 2011 May;118(5):773-81. doi: 10.1007/s00702-011-0622-9. Epub 2011 Apr 3. PMID 21461962
- [Background] Ellgring H, Seiler S, Perleth B, Frings W, Gasser T, Oertel W. Psychosocial aspects of Parkinson's disease. Neurology. 1993 Dec;43(12 Suppl 6):S41-4. PMID 8264910
- [Background] Barichella M, Cereda E, Pezzoli G. Major nutritional issues in the management of Parkinson's disease. Mov Disord. 2009 Oct 15;24(13):1881-92. doi: 10.1002/mds.22705. PMID 19691125
- [Background] Joanna Briggs Institute. The Joanna Briggs Institute Best Practice Information Sheet: music as an intervention in hospitals. Nurs Health Sci. 2011 Mar;13(1):99-102. doi: 10.1111/j.1442-2018.2011.00583.x. PMID 21426462
- [Background] Marwick C. Leaving concert hall for clinic, therapists now test music's 'charms'. JAMA. 1996 Jan 24-31;275(4):267-8. No abstract available. PMID 8544252
- [Background] Bradt J, Dileo C, Grocke D. Music interventions for mechanically ventilated patients. Cochrane Database Syst Rev. 2010 Dec 8;(12):CD006902. doi: 10.1002/14651858.CD006902.pub2. PMID 21154376
- [Background] Nilsson U. The anxiety- and pain-reducing effects of music interventions: a systematic review. AORN J. 2008 Apr;87(4):780-807. doi: 10.1016/j.aorn.2007.09.013. PMID 18395022
- [Background] Glover H, Kalinowski J, Rastatter M, Stuart A. Effect of instruction to sing on stuttering frequency at normal and fast rates. Percept Mot Skills. 1996 Oct;83(2):511-22. doi: 10.2466/pms.1996.83.2.511. PMID 8902026